CLINICAL TRIAL: NCT00164515
Title: Personalized Exercise Programme (PEP) I: Physician Referral Approach to Increasing Awareness and Sustainability of Physical Activity for Overweight Adults With Mobility Limitations.
Brief Title: Increasing Physical Activity Among Overweight Women With Mobility Disabilities.
Acronym: PEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Illinois, Center on Health Promotion Research for Persons with Disabilities (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCBDDD-R04CCR523275; R04CCR518810 (Other Grant/Funding Number: CDC/NCBDDD/DHDD)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: obesity, mobility limitations, women, physical activity
MeSH Terms: conditions — Obesity; Mobility Limitation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Physical activity awareness (No Intervention): The awareness group received a physician-recommendation to exercise an informational brochure, and pedometer.
- Arm 2: Lower Support (Experimental): The lower support group received arm 1 plus monthly newsletter, weekly personalized exercise support via telephone.
  Interventions: Behavioral: Personalized exercise programme (PEP)
- Arm 3: Higher support (Experimental): The higher support group received arm 1 plus arm 2 plus a face-to-face monthly exercise support group.
  Interventions: Behavioral: Personalized exercise programme (PEP)

INTERVENTIONS:
Behavioral: Personalized exercise programme (PEP) — Physician referred overweight and obese clients to 24 month personalized exercise programme at the U. of Illinois, Chicago
  Other Names: PEP
  Arms: Arm 2: Lower Support; Arm 3: Higher support

SUMMARY:
This study aims to increase physical activity among overweight African-American women with mobility limitations.

DETAILED DESCRIPTION:
Regular, sustainable physical activity can have a dramatic effect on reducing obesity and other secondary conditions and increasing quality of life. People with mobility limitations have a higher level of physical inactivity resulting from numerous personal and environmental barriers to physical activity participation. This project will evaluate the feasibility of increasing physical activity among overweight individuals with mobility limitations through physician-referrals to a personalized exercise programme at the Chicago-based National Center on Physical Activity and Disability (NCPAD).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Self-reported mobility limitation
* BMI greater than or equal to 27
* Receiving care at the University of Illinois, Chicago (UIC) Medical Center
* Sedentary

Exclusion Criteria:

* did not receive physician approval to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Physical activity | 24 months
  Physical activity was assessed using the Physical Activity and Disability Scale (PADS), the Barriers to Physical Activity and Disbility Scale (B-PADS), (Rimmer et al 2000) and the Mobility Limitation score (Velozo et al 1999).
Body mass index (BMI) | 24 months
  Derived emperically
Blood lipids | 24 months
  Derived emperically
Weight | 24 months
  Derived emperically
Blood Pressure | 24 months
  Dervied emperically

SECONDARY OUTCOMES:
Psychosocial Health | 24 months
  Confirmed using the Quality of Wellbeing scale (Anderson et al 1989), and CARDIA-2 scale, an 11-item assessment (Allen et al 2001).

CONTACTS AND LOCATIONS:
Overall Officials: James Rimmer, Ph.D., Principal Investigator — UIChicago
Locations (1):
- University of Illinois, Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Rimmer JH, Rauworth A, Wang E, Heckerling PS, Gerber BS. A randomized controlled trial to increase physical activity and reduce obesity in a predominantly African American group of women with mobility disabilities and severe obesity. Prev Med. 2009 May;48(5):473-9. doi: 10.1016/j.ypmed.2009.02.008. PMID 19459233